CLINICAL TRIAL: NCT02314390
Title: Group- Versus Individual-Mindfulness-Based Cognitive Therapy for Patients With a Chronic Somatic Disease and Comorbid Depressive Symptoms: a Randomized Trial
Brief Title: Group- Versus Individual-Mindfulness-Based Cognitive Therapy: a Randomized Trial
Acronym: G/I-MBCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: University of Groningen (Other)
Responsible Party: Principal Investigator, Maya Schroevers, PhD, University Medical Center Groningen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FVHH
Record Dates: First submitted 2014-12-01; First posted 2014-12-11 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Depressive Symptoms
Keywords: Depression; Mindfulness; MBCT
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- G-MBCT (Experimental): Group-Mindfulness-Based Cognitive Therapy
  Interventions: Behavioral: Group-Mindfulness-Based Cognitive Therapy
- I-MBCT (Experimental): Individual-Mindfulness-Based Cognitive Therapy
  Interventions: Behavioral: Individual-Mindfulness-Based Cognitive Therapy

INTERVENTIONS:
Behavioral: Group-Mindfulness-Based Cognitive Therapy — The intervention consists of 8 weekly sessions of MBCT. Each session will be administered in a group and will last 2 1/2 hours.
  Other Names: G-MBCT
  Arms: G-MBCT
Behavioral: Individual-Mindfulness-Based Cognitive Therapy — The intervention consists of 8 weekly sessions of MBCT. Each session will be administered individually and will last 45 to 60 minutes.
  Other Names: I-MBCT
  Arms: I-MBCT

SUMMARY:
The purpose of this study is to determine whether both group and individual mindfulness-based cognitive therapy (MBCT) are effective in reducing depressive symptoms in patients with a chronic somatic disease.

DETAILED DESCRIPTION:
Depression is a common co-morbidity in patients with a chronic somatic disease which has a negative impact on patients' physical and mental health. In recent years, Mindfulness-Based Cognitive Therapy (MBCT) has gained interest and popularity as a treatment not only for preventing recurrence of depression, but also to treat current symptoms. Usually, the training is delivered in group format, thus little is known about the feasibility and effectiveness of MBCT as an individual training.

This pilot study aims to compare the effectiveness and feasibility of group and individual MBCT in reducing depressive symptoms in patients with a chronic somatic disease.

ELIGIBILITY:
Inclusion Criteria:

* Chronic somatic disease
* Age ≥ 18 and ≤ 70
* Depressive symptoms as assessed by BDI-II score ≥ 14 (cut-off score indicating the presence of at least mild symptoms of depression)

Exclusion Criteria:

* Not being able to read and write Dutch
* Severe (psychiatric) co-morbidity
* Acute suicidal ideations or behavior
* Receiving an alternative psychological treatment during or less than two months prior to starting the participation in the study

Using an antidepressant drug during participation in the present study is allowed, on condition that a patient has been on stable medication regimen for at least two months prior to inclusion in the study, and that no new treatment with an antidepressant is initiated during the course of the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2013-09; Primary Completion 2014-03 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Change in severity of depressive symptoms | Pre-treatment to post-treatment (primary measurement point; approximately 3 months after pre-treatment) and 3-months follow-up
  Severity of depressive symptoms are assessed with the Beck Depression Inventory-II

SECONDARY OUTCOMES:
Change in well-being | Pre-treatment to post-treatment (primary measurement point; approximately 3 months after pre-treatment) and 3-months follow-up
  Well-being is measured by the Well-being Index (WHO-5)
Change in generalized anxiety | Pre-treatment to post-treatment (primary measurement point; approximately 3 months after pre-treatment) and 3-months follow-up
  Generalized anxiety is measured by the Generalised Anxiety Disorder Assessment (GAD 7)

OTHER OUTCOMES:
Change in mindfulness | Pre-treatment to post-treatment (primary measurement point; approximately 3 months after pre-treatment) and 3-months follow-up
  Mindfulness is assessed with the Five Facet Mindfulness Questionnaire (FFMQ)
Change in self-compassion | Pre-treatment to post-treatment (primary measurement point; approximately 3 months after pre-treatment) and 3-months follow-up
  Self-compassion is assessed with the 12 item Self-Compassion Scales

CONTACTS AND LOCATIONS:
Overall Officials: Robbert Sanderman, Prof., Study Chair — University Medical Center Groningen